CLINICAL TRIAL: NCT04590989
Title: PREVENTOMICS: Empowering Consumers to 'PREVENT' Diet-related Diseases Through 'OMICS' Sciences - Danish Intervention Study
Brief Title: Empowering Consumers to 'PREVENT' Diet-related Diseases Through 'OMICS' Sciences
Acronym: PREVENTOMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Fundació Eurecat (Other); Simple Feast (Unknown); Alimentómica (Unknown); University of Parma (Other); ONMI (Unknown)
Responsible Party: Principal Investigator, Mads Fiil Hjorth, Associate Professor, Head of Obesity Research Section, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-361
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Overweight; Obesity; Metabolic Syndrome
Keywords: Nutrigenomics; Nutrigenetics; Metabolomics; Microbiome; Precision nutrition; Personalized nutrition; Weight management; Body weight; Obesity
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Body Weight

STUDY DESIGN:
Intervention Model Description: Eurecat will grant Simple feast and ONMI access to users' profile via PREVENTOMICS Platform in order to know which group the subject is assigned to and intervene accordingly. The profile includes the assigned group/cluster along with nutritional recommendations of each subject.
  100 individuals will be randomly assigned to one of the two intervention groups. Both groups will receive meals and recipes from Simple Feast. The control group (50 subjects) will receive meals based on general dietary recommendations whereas the meals of the personalized plan group (50 subjects) are personalized based on an analysis of their metabolic biomarkers, genetics, preferences, health status, and lifestyle habits.
  In addition, ONMI will deliver a personally tailored and actionable behavior change program (Do-Omics) to the personalized plan group while the control group will receive general advice.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomly allocated to either intervention group (personalized plan) or control group prior to commencement of the trial. The allocation will be computer generated, and stratified by metabolic clusters (oxidative stress; inflammation; carbohydrate metabolism; lipid metabolism; microbiota-generated metabolites) in a 1:1 randomization between control and intervention groups. The person responsible for generating the code will not take part in the inclusion and examination of study participants. Study staff at UCPH and participants will be blinded to the treatment group and analyses of results will be performed in a blinded fashion. Moreover, the statistical analyses of the main outcome variable will be done without breaking the code for the intervention treatment, before the primary analyses are finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Plan (PP) (Experimental): Each subject in the PP group will be allocated to one of five clusters based on their metabolic and genetic health biomarkers from samples of urine, plasma, serum, and saliva. 58 biomarkers will be included to characterize the 5 metabolic clusters/processes in the PREVENTOMICS platform: 1) oxidative stress; 2) inflammation; 3) carbohydrate metabolism; 4) lipid metabolism; 5) microbiota-generated metabolites. Eurecat Nutrition Team has prepared a list of recommended food items to increase and food to exclude/limit from the diet for each cluster. The list will be adopted by Simple Feast in creating five different menus that will encompass the 12 meals/week of breakfasts and dinners for the five different metabolic clusters. Additionally, subjects will receive personalized actionable "Do's" push notifications by ONMI. The messages are personalized based on user reports from the behavioral questionnaire at V2 in addition to inputs from the nutritional recommendations of food to increase.
  Interventions: Other: Personalized Nutrition Plan
- Control Group (Placebo Comparator): Dietary intervention:
  The second group of 50 subjects will receive meals from Simple Feast, after integrating their metabolic profile and other blood biomarkers by PREVENTOMICS, which are based on the national dietary guidelines.
  Behavioral intervention:
  Subjects will also receive nudges, after filling out ONMI's behavioral questionnaire at V2, but that will not be personalized (i.e. basic information that is available online from NHS and WHO).
  Interventions: Other: Non-Personalized Nutrition Plan

INTERVENTIONS:
Other: Personalized Nutrition Plan — * Personalized breakfasts and dinners designed and cooked by Simplefeast, delivered twice a week (eaten 6 days per week) + access to Simplefeast's App for recipes of other meals not provided (i.e. lunches and Saturdays) which are designed to match the individual nutritional recommendations.
  * Personalized behavioral change program via electronic push notifications by ONMI
  Arms: Personalized Plan (PP)
Other: Non-Personalized Nutrition Plan — * Standard meals of breakfasts and dinners designed and cooked by Simple feast, based on general dietary recommendations, and delivered to participants twice a week. In addition, they will also have access to Simple feast's recipe App for other meals not provided. The recipes presented are generic, not personalized.
  * Subjects in the control group will also be enrolled in the behavioral program by ONMI, but the program will not be personalized nor based on the same behavior change methodology as in the PP group. In other words, the control group will get information more than is triggered to take actual action (i.e. general guidelines that is available from the National Health Service and World Health Organization).
  Arms: Control Group

SUMMARY:
The over-all aim of this 10-week randomized-controlled study, taking place only in Denmark, is to examine whether the PREVENTOMICS platform integrated in an e-commerce digital tool created to deliver personalized meals and dietary advices is able to produce more favorable health effects than meals based on general dietary recommendations in overweight subjects with elevated waist circumference.

DETAILED DESCRIPTION:
PREVENTOMICs project (Empowering consumers to PREVENT diet-related diseases through OMICS sciences), coordinated by Eurecat (Spain), has developed a personalized nutrition platform with a Decision Support System (DSS) tool that integrates different disease-inducing metabolic signatures with genotype and other informative information such as the characteristics of individual's behavioural traits, to correlate health status and provide personalized nutritional plan.

To demonstrate the potential for personalization of the platform, PREVENTOMICS will be validated in three different scenarios through three different organizations carrying out intervention studies with both healthy volunteers and volunteers with abdominal obesity.

The current study in Denmark will be a 10-week double-blinded randomized (1:1 randomization), placebo-controlled trial carried out with overweight/obese subjects having elevated waist circumference living in Greater Copenhagen. After the confirmation of the inclusion criteria, 100 individuals will be randomly assigned to one of the two intervention groups. Both groups will receive meals from Simple Feast following the national guidelines of macronutrient composition. The control group (n=50) will receive meals based on general dietary recommendations whereas the meals of the second group (n=50) are personalized based on metabolic biomarkers (PP group). In addition, participants of both groups will receive electronic push notifications of behavioral change messages for the purpose of general behavioral change and improving adherence to the nutritional intervention, which will be sent during the 10-week trial by ONMI. However, subjects in the PP group will receive personally tailored and actionable behavior change prompts from the predefined ONMI's program while subjects in the control group will receive it in a non-personalized fashion with standard messages.

Our hypothesis is that delivery of personalized meal/plan through the PREVENTOMICS platform integrated with e-commerce digital tool, will promote a greater reduction in fat mass and weight, as well as producing favorable changes in blood metabolic and inflammatory biomarkers compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-65 years
* Body mass index (in kg/m2) of ≥27,0 and <40,0 (overweight and class I and II obesity)
* Elevated waist circumference (Men>94,0 cm; Women>80,0 cm)
* Possess a smart mobile phone
* Able to provide written informed consent

Exclusion Criteria:

* Diagnosis of diabetes
* History or diagnosis of heart, liver or kidney disease
* Chronic diseases e.g. cancer within the past 5 years (except adequately-treated localized basal cell skin cancer)
* Use of drugs, that in the opinion of the medically responsible investigator, are likely to affect the primary outcomes of the study
* Being lactating, pregnant or planning to become pregnant within the study period
* Participation within another clinical trial
* Other blood donation during the study
* Self-reported weight change of >5 % (increase or decrease) within 2 months prior to screening.
* Having allergies or food intolerances
* No or limited access to the Internet
* Participants not able to comply with the study protocol judged by Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Change in body fat mass from baseline to week 10 will be analyzed by means of linear mixed models including sex, age and BMI at baseline as fixed effects as well as the stratification variable (cluster). | Baseline (V2) and week 10 (V3).
  Fat mass is evaluated by use of Dual X-ray absorptiometry (DXA) scans. The DXA-scan (iDXA, Lunar Radiation Co., Madison, Wisconsin, USA) is performed at V2 and V3 to calculate the difference between the two measurements.

SECONDARY OUTCOMES:
Change in body composition from baseline to week 10: visceral and subcutaneous fat, body lean mass, weight, body mass index, waist circumference | Baseline (V2) and week 10 (V3).
  Body composition is evaluated by DXA scans at V2 and V3. Body weight will be measured after the participant has voided their bladder using a calibrated digital scale. weight will be recorded in kg to the nearest 0.1 kg. Body Mass Index (BMI) is calculated by the person's weight in kilograms divided by the square of their height in meters. Waist circumference will be measured with a stretch-resistant tape at the midpoint between the lower margin of the last palpable ribs and the top of the iliac crest. It will be measured twice to the nearest 0.5 cm and thereafter an average will be calculated.
Change in lipid profile (fasting) from baseline to week 10: total, LDL and HDL cholesterol, triglycerides, atherogenic index of plasma (AIP) | Baseline (V2) and week 10 (V3).
  Fasting blood samples will obtained after an overnight fast (from food and drinks except for water) for a minimum of 8 hours prior to the blood sampling.
Change in blood glucose, insulin, HOMA-IR (fasting) from baseline to week 10 | Baseline (V2) and week 10 (V3).
  Fasting blood samples will obtained after an overnight fast (from food and drinks except for water) for a minimum of 8 hours prior to the blood sampling.
Change in inflammatory biomarkers (fasting) - CRP, IL-6, MCP1, TNFα, IL-10, soluble ICAM1, soluble CD14 from baseline to week 10 | Baseline (V2) and week 10 (V3).
  Fasting blood samples will obtained after an overnight fast (from food and drinks except for water) for a minimum of 8 hours prior to the blood sampling.
Change in adipokines (fasting) - Leptin, Adiponectin, Leptin/Adiponectin ratio from baseline to week 10 | Baseline (V2) and week 10 (V3).
  Fasting blood samples will obtained after an overnight fast (from food and drinks except for water) for a minimum of 8 hours prior to the blood sampling.
Change in blood pressure from baseline to week 10 | Baseline (V2) and week 10 (V3).
  Systolic and diastolic blood pressure and pulse will be measured using a validated automatic device on the arm after 5-10 min rest in a resting position. The measurement is taken three times with a 1 min rest in between (four times if the last two measurements deviate >5 mmHg), and the reading is recorded to the nearest 1 mmHg. A mean value of the last two readings is used. The same arm will be used for all measurements at all visits.

OTHER OUTCOMES:
Energy and macronutrient intake | Measurements visit (V1) and week 10 (V3).
  Validated e-FORM Food frequency questionnaire (FFQ) will be completed at visit 1 and 3. In addition, The participants are asked to fill out a complete record of everything they eat and drink (date, time, description of foods and amount) during the given days (before visit 1 and before visit 3). Participants will be asked to keep non-consecutive 3-day food registrations including one weekend day. The 3-day food record will be used to assess biomarkers of intake by Parma and to validate the Preventomics FFQ.
Quality of life assessment | Baseline (V2) and week 10 (V3).
  Quality of life will be assessed through two questionnaires:
  * EQ-5D: a standardized instrument for examining health-related quality of life. The instrument was developed by EuroQol Group. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  * Obesity and Weight-Loss Quality of Life Instrument (OWLQOL): an instrument which consists of 17 statements about weight-related feelings and emotions which are rated on a six-point scale that ranges from 0 ("not at all") to 6 ("a very great deal").
Physical activity and sleep patterns | In 7 days/8 nights post visit 1 and 7 days/8 nights during the 10-week study (between V2 and V3).
  Will be measured by an accelerometer (ActiGraph GT3X+). Participants will also have to complete a log sheet to assess bed times as well as times of removing and replacing the monitor 'ActiGraph' for the 8 nights the accelerometer is used.
Stress assessment | Baseline (V2) and week 10 (V3).
  Stress assessment will be conducted through the perceived stress scale (PSS). It is one of the most widely used psychological instruments. It measures the degree to which participants perceive events in their life as being stressful. The PSS asks about thoughts and feelings over the last month using a response scale from 0 (never) to 4 (very often).
Eating behavior | Baseline (V2) and week 10 (V3).
  Eating behavioral assessment will be done by administrating the three factor-eating questionnaire (TFEQ). It is a 51-item self-report questionnaire. The instrument measures three domains of eating behavior: (1) 'cognitive restraint of eating', (2) 'disinhibition' and (3) 'hunger'.
Attitude to weight management diets | Baseline (V2) and week 10 (V3).
  Via Diet Satisfaction Questionnaire (DSat-28) that involves 28 statements grouped into 5-scales (healthy lifestyle, eating out, cost, preoccupation with food, and planning and preparation) to evaluate individual's satisfaction with weight-management diets.
Money expended on food per household | Baseline (V2) and week 10 (V3).
  two questions will be asked in regard to the amount of money expended on food per household.
Liver and renal health markers (ALT, GGT, Uric acid, Creatinine) | Baseline (V2) and week 10 (V3).
  Fasting blood samples will obtained after an overnight fast (from food and drinks except for water) for a minimum of 8 hours prior to the blood sampling.
Microbiota composition | Baseline (V2) and week 10 (V3).
  One collection of feces will be performed within 24 hours prior to the clinical investigation day (V2 and V3). Samples will be collected and stored for future analysis. Baseline composition [eg. Enterotype] as diet-specific predictor of weight/fat loss and diet-specific change in compostion from baseline to week 10.
Urine and blood metabolome | Baseline (V2) and week 10 (V3).
  Urine spot samples and blood samples will be obtained on the intervention days (V2 and V3). The samples will be stored for future metabolomics analysis. Baseline composition [e.g. a defined number of metabolites] as a diet-specific predictor of weight/fat loss and diet-specific change in compostion from baseline to week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Mads F Hjorth, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Firstly, the IPD are to be shared within the PREVENTOMICS concortium. Secondly, the IPD will be made available upon request pending approval of a research proposal and statistical analysis plan and execution of a data sharing/prosessing agreement (according to GDPR).
  Thirdly, the IPD will be made publically available for everyone once it is completely anonymised which is 5-10 years after completion of the study (according to GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Firstly, the IPD are to be shared within the PREVENTOMICS concortium [Time Frame: Just after study completion].
  Secondly, the IPD will be made available upon request pending approval of a research proposal and statistical analysis plan and execution of a data sharing/prosessing agreement (according to GDPR) [Time Frame: After publication of primary outcome and until 5-10 years after completion of study].
  Thirdly, the IPD will be made publically available for everyone once it is completely anonymised which is 5-10 years after completion of the study (according to GDPR) [Time Frame: from 5-10 years after completion and forward] .
Access Criteria: See above

REFERENCES:
- [Derived] Galekop MMJ, Uyl-de Groot C, Redekop WK. Economic Evaluation of a Personalized Nutrition Plan Based on Omic Sciences Versus a General Nutrition Plan in Adults with Overweight and Obesity: A Modeling Study Based on Trial Data in Denmark. Pharmacoecon Open. 2024 Mar;8(2):313-331. doi: 10.1007/s41669-023-00461-8. Epub 2023 Dec 19. PMID 38113009
- [Derived] Aldubayan MA, Mao X, Laursen MF, Pigsborg K, Christensen LH, Roager HM, Nielsen DS, Hjorth MF, Magkos F. Supplementation with inulin-type fructans affects gut microbiota and attenuates some of the cardiometabolic benefits of a plant-based diet in individuals with overweight or obesity. Front Nutr. 2023 Apr 25;10:1108088. doi: 10.3389/fnut.2023.1108088. eCollection 2023. PMID 37181156
- [Derived] Aldubayan MA, Pigsborg K, Gormsen SMO, Serra F, Palou M, Galmes S, Palou-March A, Favari C, Wetzels M, Calleja A, Rodriguez Gomez MA, Castellnou MG, Caimari A, Galofre M, Sunol D, Escote X, Alcaide-Hidalgo JM, M Del Bas J, Gutierrez B, Krarup T, Hjorth MF, Magkos F. A double-blinded, randomized, parallel intervention to evaluate biomarker-based nutrition plans for weight loss: The PREVENTOMICS study. Clin Nutr. 2022 Aug;41(8):1834-1844. doi: 10.1016/j.clnu.2022.06.032. Epub 2022 Jun 30. PMID 35839545
- [Derived] Aldubayan MA, Pigsborg K, Gormsen SMO, Serra F, Palou M, Mena P, Wetzels M, Calleja A, Caimari A, Del Bas J, Gutierrez B, Magkos F, Hjorth MF. Empowering consumers to PREVENT diet-related diseases through OMICS sciences (PREVENTOMICS): protocol for a parallel double-blinded randomised intervention trial to investigate biomarker-based nutrition plans for weight loss. BMJ Open. 2022 Mar 29;12(3):e051285. doi: 10.1136/bmjopen-2021-051285. PMID 35351696